CLINICAL TRIAL: NCT05339516
Title: The Association Between Urinary Incontinence, Physical Performance and Physical Activity Level in Women With Low Back Pain a Cross-Sectional Study
Brief Title: The Association Between Urinary Incontinence, Physical Performance, Physical Activity Levels in Women With Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pinar Yasar (Other)
Responsible Party: Sponsor-Investigator, Pinar Yasar, Research Assistant, Physiotherapist, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Other Study IDs: 72867572-050.01.04-
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain; Physical Inactivity; Urinary Incontinence
MeSH Terms: conditions — Low Back Pain; Sedentary Behavior; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group
- Women with low back pain

SUMMARY:
The study is searching for the correlation between low back pain(LBP), physical performance, urinary incontinence and physical activity levels in women. Lower physical performance, more frequent urinary incontinence and less physical activity are expected in women who have LBP.

ELIGIBILITY:
Inclusion Criteria For Healthy Group:

* 30-65 years women
* Agreeing to involve in the study

Inclusion Criteria For Women With Low Back Pain Group:

* 30-65 years women
* Having low back pain for at least 3 months
* Scoring pain at least 1 in Visual Analog Scale(VAS)
* Agreeing to involve in the study

Exclusion Criteria:

* Any kind of surgery history in low back area
* Surgery history in lower limbs
* Acute low back pain
* Having a neurological disease
* Having sensory deficists
* The ones with rheumatological diseases which can cause low back pain
* Being pregnant
* Having a disc hernia pressuring to sacral nerves

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30-65 ages women who live in city of Isparta in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale(VAS) | Baseline
  Visual Analogue Scale (VAS) will be used to evaluate the severity of low back pain. The back pain they feel during activity and rest will be questioned separately from the participants. For this assessment, patients will be asked to mark their pain intensity on a 10-centimeter line. Pain intensity will be determined by measuring the distance of the marked point to the "0" point with a tape measure. Scoring is made between 0-10 and "0 means no pain"- "10 means the most severe pain imaginable".
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Baseline
  The six-question form allows evaluation of the frequency of urinary incontinence and during which activities it occurs. The validity and reliability study of the Turkish version of the test was done by Çetinel et al. made by Scoring is done with frequency, amount and degree of impact questions, a total score between 0-21 is obtained. A low score indicates that urinary incontinence affects the quality of life less, and a high score indicates that the involvement is high. For the ICIQ-SF, a score of 8 and above was determined as the most appropriate cut-off value for irritating urine leakage.
International Physical Activity Questionnaire(IPAQ) | Baseline
  The physical activity level of the participants will be evaluated with the International Physical Activity Questionnaire (IPAQ). The survey consists of a total of 5 sections and 27 questions. Information is obtained about the light, moderate and vigorous activities that the person has done in the last week and the sitting time. For physical activities performed for at least 10 minutes, the MET value (metabolic equivalent) is multiplied by the number of days and minutes to obtain the MET-min/week score. Classification according to the energy level spent in METs is made as no physical activity (MET=<600), insufficient activity (MET=600-3000), and adequate activity level (MET= >3000).
Muscle Strength Testing | Baseline
  The muscle strength of the participants will be determined by the Manual Muscle Test. The person is asked to move against gravity by taking the appropriate position for the muscle to be evaluated. If the movement can be done up to the desired part (3) it is scored as medium, if it receives minimal resistance (3+) if it gets a little good from the middle, if it can get moderate resistance (4) good, if it can get full resistance (5) it is normal. Muscle strength of the shoulder and elbow flexors in the upper extremity and hip flexors in the lower extremities will be evaluated.
Endurance Testing | Baseline
  Trunk Flexor Endurance test and Wall-Sit-Hold Test will be used to evaluate trunk and lower extremity endurance.
  Wall-Sit- Hold Test: The participant leans his back against the wall, spreads his feet shoulder-width apart and squats by bringing his knees to 90 degrees of flexion. The time during which the position can be held is recorded
Agility Testing | Baseline
  Burpee Agility Test will be used for the agility evaluation of the participants. The test consists of 4 stages. Initially, the standing participant moves into a half-squat position, then into a stance on the floor with hands and feet close together. Then the participant takes the plank position with the arms fully extended by throwing his legs back and then returning to the previous position. He then stands up and returns to the starting position and claps his hands above his head once. The standard test duration is 3 minutes, but a modified version of 1 minute will be used in order to be applicable to individuals with low physical activity.
Flexibility Testing | Baseline
  Flexibility will be assessed with the sit and reach test. The person sits in a long sitting position with his legs straight, the soles of the feet are in contact with the 31 cm high evaluation table. The participant is then asked to reach forward as far as he can, keeping his knees straight, with one hand on the other. Starting position and the farthest point that the middle finger can reach at the end of the movement is measured and the difference is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Isparta, Turkey (Türkiye)